CLINICAL TRIAL: NCT05177471
Title: Efficacy and Safety of JAK Inhibitors in Patients With Systemic Sclerosis and Interstitial Lung Disease
Brief Title: Efficacy and Safety of JAK Inhibitors in Systemic Sclerosis-associated Interstitial Lung Disease
Acronym: SCLEROJAKI
Status: Withdrawn | Type: Observational
Why Stopped: no eligible patients
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Paul DECKER, MD, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2021PI233
Record Dates: First submitted 2021-12-15; First posted 2022-01-04 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Systemic Sclerosis; Interstitial Lung Disease
MeSH Terms: conditions — Scleroderma, Systemic; Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SSc-ILD patients with JAK inhibitors

SUMMARY:
Systemic sclerosis (SSc) is a heterogeneous systemic autoimmune disease with distinct prognosis according to patients. In patients with systemic sclerosis, interstitial lung disease (ILD) concerns almost 50 % of patients and represents the main cause of mortality.

Janus kinases (JAK) inhibitors are recent therapies in the field of systemic autoimmune diseases, already approved in patients with rheumatoid arthritis.

Use of JAK inhibitors in systemic sclerosis is based on their anti-inflammatory and anti-fibrotic properties. Several preclinical murine models of systemic sclerosis demonstrated the efficacy of ruxolitinib and tofacitinib on cutaneous and pulmonary fibrosis. Recently, tofacitinib was evaluated in SSc patients in two clinical studies and showed significant improvement on skin fibrosis.

The objective of this study is to evaluate efficacy and safety of JAK inhibitors in SSc patients with ILD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with systemic sclerosis according to 2013 ACR/EULAR criteria
* Patients with interstitial lung disease affecting at least 10 % of the lungs on HRCT chest, FVC of at least 40 % of the predicted value and DLCO between 30 % and 90 % of the predicted value
* Use of JAK inhibitors

Exclusion Criteria:

* Patients with an alternative diagnosis of SSc-associated ILD (silicosis, sarcoidosis, lung cancer or other significant lung abnormalities)
* Patients with pulmonary arterial hypertension defined on right heart catheterization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with systemic sclerosis-interstitial lung disease
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2024-08-26 (Actual)

PRIMARY OUTCOMES:
relative change in FVC after 12 months of JAK inhibitor | at JAK inhibitor initiation (J0) and 12 months after JAK inhibitor initiation
  relative change in %predicted FVC after 12 months of JAK inhibitor

SECONDARY OUTCOMES:
relative change in DLCO after 12 months of JAK inhibitor | at JAK inhibitor initiation (J0) and 12 months after JAK inhibitor initiation
  relative change in %predicted DLCO after 12 months of JAK inhibitor
relative change in skin fibrosis after 12 months of JAK inhibitor | at JAK inhibitor initiation (J0) and 12 months after JAK inhibitor initiation
  relative change in modified Rodnan skin score after 12 months of JAK inhibitor

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nancy, Vandœuvre-lès-Nancy, Grand Est, France